CLINICAL TRIAL: NCT03422354
Title: Effect of Ultrasound Guided L1,L2 Paravertebral Block in Decrease the Requirements for Hypotensive Drugs During General Anesthesia in Patients Undergoing Hip Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Hala Mostafa Gomaa (Unknown); Abdelhamid, Bassant Mohamed, M.D. (Individual); Mohamed saeid Ali (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N -73/2017
Record Dates: First submitted 2017-12-27; First posted 2018-02-05 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Ultrasound Guided L1,L2 Paravertebral Block
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: after approval of the ethical committee (N-73-2017)Which approval date was 12/2/2018 74 patients scheduled for elective hip surgery were included in the study after detailed description and signing a detailed informative consent (figure1). The patients were randomized to two groups using a computer-generated list and kept in a sealed envelope into two groups:
  * Group P: 37 patients were received single shot L1-L2 paravertebral block before undergoing general anesthesia (GA).
  * Group G: 37 patients were received GA. The target of the mean blood pressure was to be more than 50mm Hg while the systolic pressure to be between 80 and 100 mm Hg and the diastolic blood pressure targeted to be 50 to 70 mmHg.
Who Masked: Care Provider, Investigator
Masking Description: The patients were randomized to two groups using a computer-generated list and kept in a sealed envelope into two groups:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block Group (Active Comparator): Patients will receive single shot L1-L2 PVB before undergoing GA Full monitoring with ECG , NIBP , puls oximetry will be applied. The level between L1 and L2 will be identified using U/S as well as transverse processes depth. Insertion points will be marked 2.5 cm lateral to the superior aspect of corresponding spinous processes, A 22-gauge Tuohy needle will be advanced until it made contact with the transverse process. The needle will be withdrawn slightly and walked off caudally to an additional depth of 1 cm. Once this is reached, 20cc of bupivacaine 0.25% will be injected slowly To control intraoperative blood pressure, fentanyl will be used as well as hypotensive drugs ( propranolol and nitroglycerine and the total dose will be recorded.
  Interventions: Procedure: Ultrasound guided PVB with General Aneasthesia; Device: Ultrasound; Drug: Paravertebral block; Drug: General Aneasthesia
- General anesthesia Group (Active Comparator): Patients will receive only GA All patients in the study will receive GA in the form of propofol 2mg/kg , atracurium 0.5ml/kg ,fentanyl 100 microgram in induction with ETT and mechanical ventilation , full monitoring with ECG , NIBP and puls oximetry will be applied.
  To control intraoperative BP,fentanyl will be used as well as,hypotensive drugs ( propranolol and nitroglycerine and the total dose will be recorded.
  To achieve post operative analgesia, intravenous paracetamol( 1gram ) and pethidine IV (50 mg ) will be added when needed
  Interventions: Device: Ultrasound; Drug: General Aneasthesia

INTERVENTIONS:
Procedure: Ultrasound guided PVB with General Aneasthesia — An 18G Tuohy needle was inserted perpendicularly at L1,2 to hit the transverse process via an out-of-plane approach. This then directed over the top of the bony structure. The deviation of the needle was kept at 15°. The space was identified using loss of resistance without U/S After negative aspiration, Transverse process visualisation was possible. Distances measured using U/S correlated well with needle depth. Injection of local anaesthetic was visualised as turbulence at L1,2 in all patients. The onset time for this block is 15-25 min
  Arms: Paravertebral block Group
Device: Ultrasound — Ultrasound
Drug: Paravertebral block — Patients will receive single shot L1-L2 PVB before undergoing GA
  Arms: Paravertebral block Group
Drug: General Aneasthesia — General Aneasthesia

SUMMARY:
The paravertebral block (PVB) is a block of the mixed nerve soon after it exits the intervertebral foramen.(2) It provides intense unilateral analgesia of long duration and has become the primary anesthetic for many applications.(3) Paravertebral Block (PVB) involves injection of local anaesthetic in a space immediately lateral to where the spinal nerves emerge from the intervertebral foramina. This technique is being used increasingly for not only intra-operative and post-operative analgesia but also as a sole anaesthetic technique for carrying out various procedures. This popularity is mainly due to the ease of the technique and fewer complications.(4) The increasing demand for hip arthroplasties over the last decades has sparked the creation of new and innovative anesthetic techniques and analgesic pathways with the goal to support best possible outcomes among this frequently elderly patient population. As a result, today different perioperative treatment pathways are available to physicians and their patients. In this context, the focus has shifted to techniques based on regional anesthetic and analgesic techniques. This trajectory has been fueled by a number of advantages including effective, long-lasting and focused pain control, decreased need for systemic analgesics and earlier mobilization.

DETAILED DESCRIPTION:
Paravertebral block group: The patient will be reviewed then moved to the block area. Intravenous access, commencement of IV crystalloid, and standard patient monitoring with ECG , NIBP , pulse oximetry Sedation 2 mg midazolam and oxygen will be commenced prior to insertion of the block.

The equipments area 22-gauge, 8 cm Tuohy needle (Perifix Epidural Needle), Skin antiseptic solution, Sterile gloves, marking pen, 1-2 ml of 1% lignocaine for skin infiltration and 20 ml of 0.25% Bupivacain.

The patient will be positioned in lateral decubitus position with the side to be blocked upward and supported by an attendant. The back should assume kyphosis.

The following boney surface anatomy landmarks are helpful to identify spinal levels and to estimate the position of the transverse processes: Iliac crest (corresponds to L3-4 or L2-3), Spinous processes (midline) , Tips of scapulae (corresponds to T7), Midline and 2.5 cm lateral to the midline.

The level between L1 and L2 will be identified using ultrasound as well as transverse processes depth. Insertion points will be marked 2.5 cm lateral to the superior aspect of corresponding spinous processes, A skin wheal will be made using lidocaine 1% at each level and then a 22-gauge, 8 cm Tuohy needle (Perifix Epidural Needle) will be advanced until it made contact with the transverse process. The needle will be withdrawn slightly and walked off caudally to an additional depth of 1 cm. Once this is reached, 20cc of bupivacaine 0.25 %( 10ml for each level) will be injected slowly after negative aspiration was confirmed at each level.

An 8-14 MHz curved array probe (Siemens ACUSON X300 Ultrasound System) was applied longitudinally to the paravertebral area.

An 18G Tuohy needle was inserted perpendicularly at L1,2 to hit the transverse process via an out-of-plane approach. This was then directed over the top of the bony structure. The deviation of the needle from the perpendicular line was kept at 15°. The paravertebral space was identified using loss of resistance to normal saline injection without ultrasound. After negative aspiration, Transverse process visualisation was possible. Distances measured using ultrasound correlated well with needle depth. Injection of local anaesthetic was visualised as turbulence at L1,2 in all patients. Ultrasound imaging not only helped determine needle insertion sites, but also provides information on the depth to the paravertebral space.

The onset time for this block is 15-25 min. The first sign of the blockade is the loss of pin-prick sensation at the dermatomal distribution of the L1 and L2 roots.

After finishing the block the patient will be moved to the operation room.

All patients in the study will receive general anesthesia in the form of propofol 2mg/kg , atracurium0.5ml/kg ,fentanyl 100 microgram in induction with ETT and mechanical ventilation , full monitoring with ECG , NIBP , puls oximetry will be applied.

To control intraoperative blood pressure, fentanyl will be used as well as, hypotensive drugs ( propranolol and nitroglycerineand the total dose will be recorded.

To achieve post operative analgesia, intravenous paracetamol( 1gram ) and pethidine IV (50 mg ) will be added when needed.

All the doses of the drugs intraoperative and postoperative will be collected.

After completion of surgical procedure and emergence from anesthesia the patient will be referred to the recovery then will be discharged to ward unit by request of surgeon for close observation.

Hemodynamics will be recorded; requirements for opioids and hypotensive drugs will be recorded and observing postoperative pain and postoperative analgesic requirements.

Pain assessment by the aid of Visual analogue scale (VAS), which is consisted of a "10 cm" line with one end labeled no pain and other end labeled worst intolerable pain. The patients marked the line at the point that best describing the pain intensity. The preoperative assessment included training of the patients about (VAS) for postoperative pain. The length of the line to the patient's mark will be measured and recorded postoperative after 30 min., 2,4, 6, 8,12 and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

Patients from 20 to 60 years.

* Genders eligible for study: both.
* ASA I-II.
* No contraindications for application of regional anesthesia as Patient refusal, local anesthetic, allergy, local sepsis or infection at puncture site, INR > 1.5 or < 12 hours post LMWH.

Exclusion Criteria:

1. Extremes of age.
2. ASA III-IV.
3. Hypovolemia.
4. Increased intracranial pressure.
5. Coagulopathy or thrombocytopenia less than 100000/ml.
6. Sepsis (increased risk of meningitis).
7. Infection at the puncture site.
8. Pre-existing neurologic disease.
9. Patient refusal.
10. History of allergy to local anesthetic.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Dose of hypotensive drugs | One day postoperatively
  Required dose of hypotensive drugs in both groups

SECONDARY OUTCOMES:
Pain assessment | One day postoperatively
  Pain assessment by the aid of Visual analogue scale (VAS)
Total dose of opioids | One day postoperatively
  Any additional analgesia during the 1st 24 hours will be covered by paracetamol 1000 mg IV infusion slowly on 10 minutes according to the patient's request. After 24 hours the total doses will be calculated

OTHER OUTCOMES:
Blood transfusion recorded | One day postoperatively
  Need for intraoperative blood transfusion will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate